## Statistical Analysis Plan Uterotonic prophylaxis after D&E

PI: Jennifer Kerns University of California, San Francisco

## **Statistical Analysis Plan**

We plan to use t-tests for continuous variables and a chi-square analysis for categorical variables for comparison of study groups at baseline. In the event that the groups are not comparable at baseline, we will do a multivariable analysis adjusting for possible confounders. We will do an intent-to-treat analysis as our primary analysis. If a woman is noted to have elevated blood pressure (>140/90) at the completion of the D&E, the study drug will be withheld as this would be a contraindication for MM. These women will still be analyzed in their original randomization group to ensure fidelity to randomization's goal of balancing confounders. In addition to computing the dichotomous outcome of blood loss > 125cc and/or intervention for bleeding, we will also compare the number of interventions listed in Table 1 for each group. We will also do a sensitivity analysis of the composite outcome in which we exclude the more minor interventions for bleeding, use of uterotonics or manual pressure. For our secondary outcome of mean blood loss difference, we will also conduct a per-protocol analysis, comparing those who received any uterotonic medication (placebo plus additional doses as well as intervention arm plus or minus additional doses) versus those who received no utertonic.

Version: April 10 2014